CLINICAL TRIAL: NCT07237620
Title: Comparison of Calcium Hydroxide and Diclofenac Sodium as Intracanal Medicaments on Periapical Healing: A Fractal Analysis Study
Brief Title: The Effect of Different Intracanal Medicaments on Periapical Lesion Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Merve Sari, Assistant Professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1109202503
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Periapical Lesion Healing; Apical Periodontitis
Keywords: Apical Periodontitis; intracanal medicaments; Diclofenac sodium; Calcium hydroxide; Fractal analysis; Endodontic retreatment
MeSH Terms: conditions — Periapical Periodontitis | interventions — Diclofenac; Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, parallel-group, double-blind, randomized controlled clinical trial.
Who Masked: Participant, Investigator
Masking Description: Patients are to be randomly assigned into two groups (Ca(OH)₂ and DCS) using a four-block randomization technique (allocation ratio 1:1) via www.randomizer.org. The intracanal medicaments are to be prepared by an independent clinician not involved in the study. Both the operator and the patient are to be blinded to the type of medicament used. The medicaments will have similar appearance, color, and consistency to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diclofenac sodium (Experimental): 1 g of DCS (Fagron, Rotterdam, Netherlands) is to be mixed with 1 mL of distilled water.
  After preparation, the medicaments are to be placed into the canal using a size 25 lentulo spiral (Dentsply Sirona, Switzerland) set 2 mm short of the working length. The medicament is to be condensed to the canal orifice with a sterile paper point.
  Interventions: Procedure: Diclofenac sodium
- Calcium hydroxide (Active Comparator): 1 g of CH (Kalsin, Konya, Turkey) is to be mixed with 1 mL of distilled water.After preparation, the medicaments are to be placed into the canal using a size 25 lentulo spiral (Dentsply Sirona, Switzerland) set 2 mm short of the working length. The medicament is to be condensed to the canal orifice with a sterile paper point.
  Interventions: Procedure: Diclofenac sodium

INTERVENTIONS:
Procedure: Diclofenac sodium — Group 1: 1 g of CH (Kalsin, Konya, Turkey) is to be mixed with 1 mL of distilled water.
  Group 2: 1 g of DCS (Fagron, Rotterdam, Netherlands) is to be mixed with 1 mL of distilled water.
  After preparation, the medicaments are to be placed into the canal using a size 25 lentulo spiral (Dentsply Sirona, Switzerland) set 2 mm short of the working length.
  Other Names: Calcium hydroxide

SUMMARY:
This study is planned to evaluate the effects of two different intracanal medicaments-calcium hydroxide and diclofenac sodium-on periapical healing following endodontic retreatment. Fifty-four patients will be included and randomly assigned into two groups according to the type of medicament used. All procedures will be performed by a single experienced endodontist under standardized clinical conditions. Periapical lesion healing will be assessed radiographically at baseline and after 12 months using fractal analysis to quantitatively evaluate bone regeneration. The primary outcome will be the change in the fractal dimension values between the initial and follow-up radiographs.

DETAILED DESCRIPTION:
Removal of Previous Root Canal Filling All stages of the root canal procedure are to be performed by a single endodontist with seven years of clinical experience. Local anesthesia is to be achieved with supraperiosteal infiltration of 4% articaine containing 1:100,000 epinephrine (Ultracain D-S; Sanofi, Paris, France). The tooth is to be isolated with a rubber dam, and canal access is to be achieved through a conventional access cavity. The filling material in the access cavity is to be removed using a water-cooled diamond fissure bur.

Root filling material is to be removed using ProTaper Universal Retreatment files operated at 500 rpm. D1 (30/0.09), D2 (25/0.08), and D3 (20/0.07) files are to be used in the coronal, middle, and apical thirds, respectively. Apical patency is to be verified, and the master apical file (MAF) is to be used up to the working length, which is to be determined when the electronic apex locator (Morita Root ZX, Tokyo, Japan) displays "0.0" and confirmed radiographically.

The MAF is to be selected according to the canal volume, and canal preparation is to be completed. Retreatment is to be considered complete when no residual filling material is observed radiographically.

Medication Application and Randomization Patients are to be randomly assigned into two groups (Ca(OH)₂ and DCS) using block randomization technique (allocation ratio 1:1) via www.randomizer.org. The intracanal medicaments are to be prepared by an independent clinician not involved in the study. Both the operator and the patient are to be blinded to the type of medicament used. The medicaments will have similar appearance, color, and consistency to maintain blinding.

Group 1: 1 g of CH (Kalsin, Konya, Turkey) is to be mixed with 1 mL of distilled water.

Group 2: 1 g of DCS (Fagron, Rotterdam, Netherlands) is to be mixed with 1 mL of distilled water.

After preparation, the medicaments are to be placed into the canal using a lentulo spiral (Dentsply Sirona, Switzerland) set 2 mm short of the working length. The medicament is to be condensed to the canal orifice with a sterile paper point. The canals are to be sealed with a sterile cotton pellet and Cavit (3M ESPE, Seefeld, Germany).

Patients are to be prescribed 400 mg ibuprofen if needed and provided with a contact number for emergency communication in case of persistent or severe pain.

Removal of Medicaments and Root Canal Filling One week later, under rubber dam isolation, the access cavity is to be reopened. The intracanal medicaments are to be removed mechanically using the MAF and irrigation with a total of 10 mL NaOCl. The final irrigation sequence is to consist of 5 mL saline, 3 mL 17% EDTA (1 minute), 5 mL saline, 5 mL 2.5% NaOCl, and a final rinse with 5 mL saline.

All canals are to be obturated using the lateral condensation technique with Bioserra sealer (Dentsply DeTrey GmbH, Konstanz, Germany). All endodontic procedures are to be performed by a single endodontist.

Follow-up and Outcome Evaluation The primary outcome is to be the reduction in periapical lesion volume, which will be assessed by fractal analysis of periapical radiographs obtained before treatment and at the 12-month follow-up. The images are to be analyzed by two blinded evaluators.

Patients are to be recalled after one year for clinical and radiographic evaluation. Clinical signs and symptoms (tenderness to percussion or palpation, pain, deep periodontal pockets, sinus tract, or swelling) are to be recorded Digital radiographs are to be obtained using the same X-ray holder, and standardized exposure settings to ensure consistent diagnostic quality.

All patients are to be invited for an additional follow-up after an average postoperative period of four years. Restorations are to be evaluated clinically and expected to remain of good quality throughout the observation period.

Fractal Analysis Baseline and one-year follow-up digital periapical radiographs of the teeth are to be obtained using a periapical radiography device equipped with standard size #2 photostimulable phosphor plates.

All analyses are to be performed by an experienced dentomaxillofacial radiologist who will be blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

The study is planned to include patients aged 18-60 years who are systemically healthy (ASA I-II), present with apical periodontitis after primary root canal treatment, and have single-rooted, root-filled mandibular teeth with a periapical index (PAI) score of ≥3.

Endodontic treatment failure is to be evaluated based on clinical and radiographic examinations. The duration of the initial endodontic treatment is to be at least four years or longer and/or the teeth are to exhibit clinical symptoms and signs. Previous root canal fillings are to be assessed for obturation quality and classified as satisfactory if they meet the following criteria: no visible voids, good condensation, and termination within 1-2 mm of the radiographic apex. If one or more of these criteria are not fulfilled, the obturation is to be classified as poor quality.

The presence of post-treatment apical periodontitis, poor obturation quality, and/or persistent or newly developed symptoms (such as spontaneous pain, tenderness to palpation or percussion) and/or sinus tract formation are to be considered as indications for retreatment.

Exclusion Criteria:

Patients with a history of psychiatric disorders, allergic reactions, or pregnancy, and those who have taken analgesics within seven days prior to treatment or antibiotics within the previous three months, are to be excluded from the study.

Teeth presenting with a periodontal pocket depth greater than 4 mm, severe coronal destruction preventing rubber dam placement, vertical root fracture, internal or external resorption, ankylosis, overfilling, open apex, or that have undergone surgical or nonsurgical retreatment after primary therapy are to be excluded. Teeth with perforation or fractured instruments are also to be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Periapical Lesion Healing | 1 year
  The primary outcome is to be the reduction in periapical lesion volume, which will be assessed by fractal analysis of periapical radiographs obtained before treatment and at the 12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Sarı, DDS,MSc, Principal Investigator — Mustafa Kemal University Hatay, Turkey
Locations (1):
- Merve Sarı, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD due to confidentiality and privacy considerations.

REFERENCES:
- [Background] Negm MM. Effect of intracanal use of nonsteroidal anti-inflammatory agents on posttreatment endodontic pain. Oral Surg Oral Med Oral Pathol. 1994 May;77(5):507-13. doi: 10.1016/0030-4220(94)90233-x. PMID 8028874
- [Background] Zhang S, Qu X, Tang H, Wang Y, Yang H, Yuan W, Yue B. Diclofenac Resensitizes Methicillin-Resistant Staphylococcus aureus to beta-Lactams and Prevents Implant Infections. Adv Sci (Weinh). 2021 May 3;8(13):2100681. doi: 10.1002/advs.202100681. eCollection 2021 Jul. PMID 34258168
- [Background] de Freitas RP, Greatti VR, Alcalde MP, Cavenago BC, Vivan RR, Duarte MA, Weckwerth AC, Weckwerth PH. Effect of the Association of Nonsteroidal Anti-inflammatory and Antibiotic Drugs on Antibiofilm Activity and pH of Calcium Hydroxide Pastes. J Endod. 2017 Jan;43(1):131-134. doi: 10.1016/j.joen.2016.09.014. Epub 2016 Dec 6. PMID 27939738
- [Background] Adl A, Motamedifar M, Malekzadeh P, Sedigh-Shams M. Disinfection of dentinal tubules with diclofenac sodium and N-Acetylcysteine compared with calcium hydroxide as intracanal medicaments against Enterococcus faecalis. Aust Endod J. 2022 Dec;48(3):386-391. doi: 10.1111/aej.12575. Epub 2021 Oct 7. PMID 34617640